CLINICAL TRIAL: NCT05814380
Title: The Comparisons of Regional Scintigraphic DPD Uptake Between Patients With Hereditary and Wild Type Cardiac Transthyretin Amyloidosis
Brief Title: The Regional Scintigraphic DPD Uptake in Cardiac Transthyretin Amyloidosis.
Acronym: AMYLOIDOZA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Katarzyna Holcman (Other)
Responsible Party: Sponsor-Investigator, Katarzyna Holcman, Principal Investigator, John Paul II Hospital, Krakow
Organization: John Paul II Hospital, Krakow (Other)
Other Study IDs: ID#57165999
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Transthyretin Amyloidosis
Keywords: transthyretin amyloidosis; SPECT
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: grade 1-3 cardiac retention of 99mTc-DPD in scintigraphy
  Interventions: Radiation: 99mTc-DPD scintigraphy; Diagnostic Test: Collection of blood samples and echocardiography
- Group 2: first-degree relative of a patient with ATTR
  Interventions: Radiation: 99mTc-DPD scintigraphy; Diagnostic Test: Collection of blood samples and echocardiography

INTERVENTIONS:
Radiation: 99mTc-DPD scintigraphy — 99mTc-DPD scintigraphy
Diagnostic Test: Collection of blood samples and echocardiography — Collection of blood samples from a peripheral vein and TTR sequencing. Transthoracic echocardiography.

SUMMARY:
Cardiac transthyretin (ATTR) amyloidosis is an infiltrative cardiomyopathy with an inexorably progressive clinical course and poor prognosis. The disease is caused by misfolding of the liver-derived precursor protein transthyretin as a result of an acquired wild-type variant (ATTRwt) or as a hereditary mutant variant (ATTRm). Application of single-photon emission computed tomography (SPECT) provides greater anatomic resolution, enabling the assessment of amyloid burden within individual left ventricle segments.This study aims to describe the pattern of regional myocardial distribution of 3,3-diphosphono-1,2-propanedicarboxylic acid (DPD) SPECT uptake among patients with ATTRwt and ATTRm. It will investigate the clinical, biochemical and echocardiographic, including left ventricle longitudinal strain profile in ATTRwt and ATTRm. Moreover, we will evaluate the presence and extent of DPD cardiac uptake among asymptomatic ATTRm variants carriers.This is a prospective multi-center observational study. The study, after obtaining prior written informed consent, will include consecutive patients who have Grade 1-3 cardiac DPD retention in scintigraphy. In addition, first-degree relatives of patients with ATTRm are going to be enrolled. Patients are going to undergo TTR gene sequencing to assess the presence of pathogenic variants associated with ATTRm. Both planar scintigraphy, SPECT and speckle-tracking echocardiography will be reviewed and interpreted using visual and quantitative approaches.

DETAILED DESCRIPTION:
Cardiac transthyretin (ATTR) amyloidosis is an infiltrative cardiomyopathy with an inexorably progressive clinical course and poor prognosis. The disease is caused by misfolding of the liver-derived precursor protein transthyretin as a result of an acquired wild-type variant (ATTRwt) or as a hereditary mutant variant (ATTRm). Application of single-photon emission computed tomography (SPECT) provides greater anatomic resolution, enabling the assessment of amyloid burden within individual left ventricle segments.

This study aims to describe the pattern of regional myocardial distribution of 3,3-diphosphono-1,2-propanedicarboxylic acid (DPD) SPECT uptake among patients with ATTRwt and ATTRm. It will investigate the clinical, biochemical and echocardiographic, including left ventricle longitudinal strain profile in ATTRwt and ATTRm. Moreover, we will evaluate the presence and extent of DPD cardiac uptake among asymptomatic ATTRm variants carriers.

This is a prospective multi-center observational study. The study, after obtaining prior written informed consent, will include consecutive patients who have Grade 1-3 cardiac DPD retention in scintigraphy. In addition, first-degree relatives of patients with ATTRm are going to be enrolled. Patients are going to undergo TTR gene sequencing to assess the presence of pathogenic variants associated with ATTRm. Both planar scintigraphy, SPECT and speckle-tracking echocardiography will be reviewed and interpreted using visual and quantitative approaches.

The collected data will be analyzed statistically to verify research hypotheses. Approval from the local Bioethical Committee will be obtained before carrying out the study. All procedures performed are going to be in accordance with the ethical standards of the 1964 Helsinki declaration and its later amendments, or comparable ethical standards.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age,
* providing written informed consent,
* grade 1-3 cardiac retention of 99mTc-DPD in scintigraphic study or a first-degree relative of a patient with ATTR

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 consecutive patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-05-04 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
regional left ventricle 99mTc-DPD uptake | day 1
  To compare the regional left ventricle 99mTc-DPD uptake among patients with hereditary and wild-type cardiac transthyretin amyloidosis.

SECONDARY OUTCOMES:
right ventricular 99mTc-DPD accumulation | day 1
  To assess prevalence of right ventricular 99mTc-DPD accumulation among patients with hereditary and wild-type cardiac transthyretin amyloidosis.
99mTc-DPD cardiac uptake among asymptomatic hereditary transthyretin amyloidosis variants carriers | day 1
  To evaluate the presence and extent of 99mTc-DPD cardiac uptake among asymptomatic hereditary transthyretin amyloidosis variants carriers.

OTHER OUTCOMES:
left ventricle longitudinal strain | day 1
  To investigate echocardiographic left ventricle longitudinal strain profile in hereditary and wild-type ATTR cardiac amyloidosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiac and Vascular Diseases, John Paul II Hospital, Krakow, Lesser Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holcman K, Rubis P, Cmiel B, Zabek A, Boczar K, Stepien-Wroniecka A, Graczyk K, Mroz K, Dziewiecka E, Mateusz W, Szczepara S, Kurek M, Gutkowska K, Podolec P, Kostkiewicz M. The left ventricular mechanical dispersion as a marker of disease severity in transthyretin cardiac amyloidosis. Sci Rep. 2025 Nov 27;15(1):42372. doi: 10.1038/s41598-025-26329-x. PMID 41309713
- [Derived] Holcman K, Rubis P, Podolec P, Ostrowska M, Stepien-Wroniecka A, Graczyk K, Mroz K, Zabek A, Boczar K, Dziewiecka E, Winiarczyk M, Cmiel B, Kurek M, Kostkiewicz M. Transthyretin-related amyloid cardiomyopathy: A single-center experience in southern Poland, an endemic area. Kardiol Pol. 2025;83(9):1039-1052. doi: 10.33963/v.phj.107207. Epub 2025 Jul 11. PMID 40643127
- [Derived] Holcman K, Rubis P, Cmiel B, Stepien A, Graczyk K, Mroz K, Szot W, Dziewiecka E, Winiarczyk M, Kurek M, Keska M, Podolec P, Kostkiewicz M. Pre-symptomatic scintigraphic and genetic cascade screening in cardiac transthyretin amyloidosis. Eur J Nucl Med Mol Imaging. 2025 Apr;52(5):1840-1852. doi: 10.1007/s00259-024-06966-6. Epub 2024 Nov 14. PMID 39537877